CLINICAL TRIAL: NCT07156968
Title: Can Different Intrathecal Drugs Affect Day Case Anal Surgery Recovery Duration?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nasser Sayed, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R 138 / 2021
Record Dates: First submitted 2024-08-26; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Effect of Drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The bupivacaine-fentanyl group (Experimental)
  Interventions: Drug: Bupivacaine-fentanyl
- The prilocaine-fentanyl group (Experimental)
  Interventions: Drug: Bupivacaine-fentanyl
- The prilocaine-dexametomidine group (Experimental)
  Interventions: Drug: Bupivacaine-fentanyl

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — A peripheral intravenous (IV) catheter will be inserted, and a 7 mL kg-1 crystalloid infusion will be initiated. The patients will be premedicated with 0.03 mg kg-1 midazolam IV. Heart rate and peripheral oxygen saturation (SpO2) will be monitored continuously; systolic, diastolic, and mean arterial pressure (MAP) will be measured noninvasively at 5 min intervals during the procedure and at 15 min intervals during the post anesthesia care unit (PACU) stay. The baseline values will be recorded. Nasal oxygen 2 L min-1 will be administered during the whole procedure
  Other Names: prilocaine-fentanyl; prilocaine-dexametomidine

SUMMARY:
This study aims to compare effect of adding fentanyl or dexmetomidine on duration of motor and sensory block after spinal anesthesia with prilocaine during day case perianal surgery and whether it impact time to discharge home.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* ASA 1-3
* height <155cm or >175cm
* Day case perianal surgery

Exclusion Criteria:

* Hypersensitivity to the study drugs
* Refusal of patients.
* Patients with contraindications for spinal anesthesia
* previous voiding difficulty
* patients taking anticholinergic medications.
* emergency cases
* Patients with contraindications for day case sitting.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Sensory block resolution to S3 block | at 1 min intervals until the maximum block will be achieved and at 15 min intervals thereafter until the block resolved to S3 dermatome.
  The sensory block will be measured at the midclavicular line with a pinprick test (via a 22 gauge hypodermic needle)
Home discharge | Home discharge will be assessed as the time from the end of surgery until the patients reach a post-anesthesia discharge score
  (modified Alderts score) ≥9, able to void spontaneously and the sensory block resolves to the S3 dermatome.
incidence of postoperative urinary retention (POUR) | within 6 hours after surgery
  The postoperative urinary retention (POUR) will be evaluated at hourly intervals in the PACU and ward; ultrasonic bladder scanning will be used for this purpose. If the bladder volume exceeds 500 mL and the patient has not voided spontaneously, urinary catheterization will be introduced.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided